CLINICAL TRIAL: NCT07323004
Title: Construction of a Motor Development Assessment System and an Improvement Mechanism for Children With Neurodevelopmental Disorders
Brief Title: Motor Development Assessment and Support for Children With Neurodevelopmental Disorders
Acronym: CAMD-NDD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aiyoudong Children and Youth Sports Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Basic-2461; 2022YFC3600204 (Other Grant/Funding Number: ministry of science and technology of the People's Republic of China)
Record Dates: First submitted 2025-04-11; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Neurodevelopmental Disorders
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- typical development (No Intervention): This group consists of typically developing children aged 4-12 years. No intervention will be applied. The group will be used as a baseline for comparison and analysis of motor development and related health fitness indicators.
- Special Intervention Group (Experimental): This group includes children aged 4-12 years diagnosed with neurodevelopmental disorders. Participants will receive a combined intervention consisting of traditional rehabilitation therapy and a structured, characteristic exercise program designed to improve motor development and core health-related fitness.
  Interventions: Behavioral: Characteristic Exercise Intervention
- General Intervention Group (Active Comparator): This group includes children aged 4-12 years diagnosed with neurodevelopmental disorders. Participants will receive standard traditional rehabilitation therapy without the additional characteristic exercise intervention.
  Interventions: Behavioral: Traditional Rehabilitation

INTERVENTIONS:
Behavioral: Characteristic Exercise Intervention — This intervention combines traditional rehabilitation techniques (e.g., occupational therapy and physical therapy focusing on fine and gross motor skills) with a structured, age-appropriate characteristic exercise program. The program includes dynamic balance training, sensory-motor integration activities, rhythmic movement games, and core stability exercises.
  * Frequency: 3 sessions per week
  * Duration: 45 minutes per session
  * Total Intervention Period: 12 weeks
  * Distinguishing Feature: The inclusion of customized play-based movement training and sensory-motor games designed specifically to support neurodevelopmental improvement in young children with motor delays.
  Arms: Special Intervention Group
Behavioral: Traditional Rehabilitation — Participants will receive conventional rehabilitation therapy, including basic motor skill exercises, postural control training, and therapist-led occupational therapy sessions aimed at improving daily motor function.
  * Frequency: 3 sessions per week
  * Duration: 45 minutes per session
  * Total Intervention Period: 12 weeks
  * Distinguishing Feature: This group receives only traditional rehabilitation techniques without any additional structured or characteristic physical activity component.
  Arms: General Intervention Group

SUMMARY:
On the one hand, it helps to understand the motor development of preschool children, so as to provide early intervention means for the prevention of motor retardation and promote the healthy development of preschool children, and on the other hand, different motor intervention strategies are formulated according to the developmental characteristics of children with different core symptoms. It is of great academic value to verify the effectiveness of the program through empirical research on exercise intervention and promote the improvement of motor and cognitive development of children with neurodevelopmental disorders.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 12 years
* Born at full term (gestational age ≥ 37 weeks and < 42 weeks)
* Provided informed consent signed by their legal guardian
* For the ADHD group:
* Diagnosed with Attention-Deficit/Hyperactivity Disorder (ADHD) by a qualified physician (e.g., child psychiatrist or psychologist) according to DSM-5 diagnostic criteria
* For the typical development (control) group:
* No symptoms related to ADHD (e.g., inattention, hyperactivity, impulsivity)
* Normal scores on parent- and teacher-rated behavioral questionnaires (e.g., CBCL, SDQ)
* No history of neurological or psychiatric disorders

Exclusion Criteria:

* Diagnosis of other neurodevelopmental disorders, such as:
* Autism Spectrum Disorder (ASD)
* Learning disabilities
* Epilepsy, cerebral palsy, or other neurological conditions
* Developmental quotient (DQ) < 85, as measured by standardized tools (e.g., Gesell scale)
* Significant visual or hearing impairments, or congenital malformations
* History of high-risk birth events, including but not limited to:
* Severe birth asphyxia
* Intrauterine infections
* Presence of genetic or metabolic disorders, or severe dysfunction of vital organs
* For the ADHD group: comorbid psychiatric conditions (e.g., schizophrenia, severe mood disorders)

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gross Motor Development | Baseline, Week 6 (midpoint), and Week 12 (post-intervention)
  Assessed using the Test of Gross Motor Development-3 (TGMD-3), which evaluates locomotor and object control skills.The scoring ranges from the lowest score of 0 to the highest score of 104 points, and the higher the score, the better the level of motor development.
Change in Motor Coordination | Baseline, Week 6, and Week 12
  Evaluated with the Movement Assessment Battery for Children-Second Edition (MABC-2), which measures manual dexterity, aiming and catching, and balance skills.
Change in Health-Related Physical Fitness | Baseline, Week 6, and Week 12
  Standing long jump (centimeters)
Change in Health-Related Physical Fitness | Baseline, Week 6, and Week 12
  Continuous two-foot jump (times)
Change in Health-Related Physical Fitness | Baseline, Week 6, and Week 12
  10m shuttle run (seconds)
Change in Health-Related Physical Fitness | Baseline, Week 6, and Week 12
  Balance Beam Walk
Change in Gross Motor Development | Baseline, Week 6 (midpoint), and Week 12 (post-intervention)
  Assessed using the Test of Gross Motor Development-3 (TGMD-3), which evaluates locomotor and object control skills.

SECONDARY OUTCOMES:
Change in gait velocity (single task condition) | Baseline and Week 12
  In single-task conditions, gait speed is measured using a plantar pressure system and reported in meters per second (m/s).
Change in step size (single-task condition) | Baseline and Week 12
  In single-task conditions, step lengths were measured using a plantar pressure system and reported in centimeters (cm).
Change in Gait Parameters and Dual-Task Cost | Baseline and Week 12
  Gait parameters under single-task condition (e.g., gait speed, step length) measured in meters/second and centimeters using a plantar pressure system.
Change in Working Memory | Baseline and Week 12
  Description: Performance on a standardized computer-based working memory task.
Change in SDNN | Baseline and Week 12
  Standard deviation of normal-to-normal intervals (SDNN) collected from ECG to assess overall heart rate variability.
Change in Gut Microbiota Composition and Inflammatory Markers（Changes in gut microbiota diversity） | Baseline and Week 12
  Diversity of gut microbiota will be analyzed by stool samples (e.g., Alpha diversity index).
Change in Gut Microbiota Composition and Inflammatory Markers(Changes in the level of the inflammatory marker IL-6) | Baseline and Week 12
  Blood samples will be analyzed for levels of the inflammatory marker interleukin-6 (IL-6), usually in picograms per milliliter (pg/mL).
Change in Gut Microbiota Composition and Inflammatory Markers(Changes in TNF-α Levels, a Marker of Inflammation) | Baseline and Week 12
  Blood samples will be analyzed for levels of the inflammatory marker tumor necrosis factor-α (TNF-α), usually in picograms per milliliter (pg/mL).
Change in Gait Parameters and Dual-Task Cost(Changes in gait speed) | Baseline and Week 12
  Gait speed is measured using a plantar pressure system and reported in meters per second (m/s) in a dual-task condition where cognitive tasks are performed.
Change in Gait Parameters and Dual-Task Cost(Changes in stride length) | Baseline and Week 12
  Under the conditions of a dual-task situation involving cognitive tasks, measure the step length using a plantar pressure system, and report the result in centimeters (cm).
Change in Gait Parameters and Dual-Task Cost | Baseline and Week 12
  Dual-task cost (percent) calculated as the relative difference between single-task and dual-task gait performance.
Change in Inhibitory Control | Baseline and Week 12
  Performance on a standardized computer-based inhibitory control task.
Change in Cognitive Flexibility | Baseline and Week 12
  Performance on a standardized computer-based cognitive flexibility task.
Change in RMSSD | Baseline and Week 12
  Root mean square of successive differences (RMSSD) collected from ECG to assess parasympathetic activity.
Change in LF/HF Ratio | Baseline and Week 12
  Low-frequency to high-frequency power ratio (LF/HF) derived from ECG spectral analysis to evaluate autonomic balance.

CONTACTS AND LOCATIONS:
Locations (1):
- China Institute of Sport Science, Beijing, China

IPD SHARING:
Plan to Share IPD: No